CLINICAL TRIAL: NCT00543153
Title: The Exceptional Patient in Cancer Care
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0435
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Exceptional Patient; Cancer Care; Interview
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with cancer
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview lasting approximately 30-45 minutes.

SUMMARY:
The objectives of this study is to conduct a multicenter, dual country (United States and Israel), study examining the experience of patients with cancer that were considered by their physicians as having exceptional course of survival related to their specific disease state.

The primary aim of the study is to develop a detailed description of patients' experience of an exceptional disease course. The secondary aim is to define the content domain for assessment and measurement of exceptional disease course in patients with cancer and identify lessons learned from these exceptional patients that can be a base for future studies to benefit others.

DETAILED DESCRIPTION:
The investigators of this study are exploring the experience of people with cancer who are considered by their physicians as having an exceptional course of disease - people who have defied the odds and remain well despite the severity of the original diagnosis.

Participation in this study is completely voluntary. Lessons learned from recorded experience(s) may be helpful to other patients and can be a basis for future studies that may benefit other patients.

To participate in this important study is simple and not time consuming. You will have only one face-to-face or telephone interview with a research assistant. During the interview you will simply be asked to describe your perspective, thoughts, and behaviors that you think are related to your disease course and lessons that you think others may gain benefit from. The interview will last about one hour and will be conducted at a time that is convenient for you.

If you agree to participate a research assistant will schedule a time for a recorded interview by phone or if possible at a location convenient to you. The interviews will be taped and transcribed. All recorded interviews will be retained for a minimum of 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ability to speak and read English with patients residing in the US, ability to speak and read Hebrew with patients residing in Israel.
3. Diagnosis of cancer confirmed by pathology.
4. Exceptional disease course as identified by patients' physician, in terms of survival and unusual disease course that is appropriately medically documented.
5. Consent to participate in this study.

Exclusion Criteria:

1. Inability to understand the intent of the study.
2. Medical condition that would preclude participation in an interview session lasting 30-45 minutes.
3. Diagnosis of active psychosis or severe cognitive impairment confirmed by the patient's attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, 18 years of age or older, dianosed with cancer that were considered by their physicians as having exceptional course of survival related to their specific disease state.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Qualitative Data Collection: Patients' Experience of Exceptional Disease Course | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Moshe A. Frenkel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- UT MD Anderson Cancer Center, Houston, Texas, United States
- Tel Aviv University, Tel Aviv, Israel

REFERENCES:
- [Result] Frenkel M, Ari SL, Engebretson J, Peterson N, Maimon Y, Cohen L, Kacen L. Activism among exceptional patients with cancer. Support Care Cancer. 2011 Aug;19(8):1125-32. doi: 10.1007/s00520-010-0918-6. Epub 2010 May 29. PMID 20512358
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org